CLINICAL TRIAL: NCT05854498
Title: Phase II Study of Liposomal Irinotecan With TAS102 and Bevacizumab for Patients With Metastatic Colorectal Cancer
Brief Title: Liposomal Irinotecan With TAS102 and Bevacizumab for Patients With Metastatic Colorectal Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-0449; Protocol Version 2/16/2024 (Other: UW Madison); UW23016 (Other: UWCCC); SMPH/MEDICINE/HEM-ONC (Other: UW Madison); NCI-2023-05190 (Registry Identifier: NCI Trial ID)
Record Dates: First submitted 2023-05-02; First posted 2023-05-11 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-04

CONDITIONS: Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — irinotecan sucrosofate; trifluridine tipiracil drug combination; Bevacizumab

STUDY DESIGN:
Intervention Model Description: This is a nonrandomized, single arm, open-label study of the combination of liposomal irinotecan with TAS102 and bevacizumab in patients with treatment refractory metastatic colorectal cancer.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Participants with Metastatic or Unresectable Colorectal Cancer (Experimental): Male and females aged 18 years and older with histologically confirmed metastatic or unresectable (not amenable to curative therapy) colorectal cancer.
  Interventions: Drug: Liposomal irinotecan; Drug: TAS102; Drug: Bevacizumab

INTERVENTIONS:
Drug: Liposomal irinotecan — 50mg/m2 IV on days 1 and 15
Drug: TAS102 — 35mg/m2 PO BID on days 1-5 and 15-19
Drug: Bevacizumab — 5mg/kg IV on days 1 and 15

SUMMARY:
This study is being done to see if combining liposomal irinotecan with TAS102 and bevacizumab confers clinical benefit for patients with treatment refractory metastatic colorectal cancer.

DETAILED DESCRIPTION:
This prospective phase II, single arm, single site trial will evaluate the efficacy of the combination of liposomal irinotecan (nal-IRI), TAS102, and bevacizumab for the treatment of patients with mismatch repair proficient, metastatic or unresectable colorectal cancer that has previously been treated with 5-fluorouracil, oxaliplatin, irinotecan and if RAS wild-type an anti-EGFR agent. A total of 25 patients will be accrued at UW Carbone Cancer Center. Subject enrollment will occur over 12 months with the total duration of the trial expected to be 3 years.

Primary Objective

* To determine the progression free survival (PFS) of patients with metastatic colorectal cancer treated in the treatment refractory setting with liposomal irinotecan in combination with TAS102 and bevacizumab.

Secondary Objectives

* To evaluate the objective response rate (ORR) of liposomal irinotecan in combination with bevacizumab and TAS102.
* To assess the safety and tolerability of these regimens in this setting.
* To determine the impact of the timing of irinotecan use in prior lines of therapy on the ORR and PFS observed with these nal-IRI containing treatment regimens

ELIGIBILITY:
Inclusion Criteria:

* Patients must be ≥ 18 years of age
* Eastern Cooperative Oncology Group (ECOG) performance must be 0 or 1.
* Patients must have a histologically or cytologically confirmed diagnosis of colorectal adenocarcinoma and be metastatic or unresectable.
* The cancer must be mismatch repair proficient.
* Patients must have had prior treatment with 5-fluorouracil, oxaliplatin, irinotecan containing regimens. If RAS wild-type must have received prior anti-EGFR therapy with either cetuximab or panitumumab. If RAS wild-type and HER2 positive then must have had a prior HER2 targeted therapy.

Exclusion Criteria:

* Uncontrolled concurrent medical illness that would not allow for the completion of the planned therapy.
* Patients whose cancers possess BRAF V600 mutations are excluded.
* Patients must stop the use of strong inducers/inhibitors of CYP3A4 at least 2 weeks before initiating therapy.
* Patients must not have mismatch repair deficient or microsatellite instability high cancers.
* Patients must not have received prior TAS102.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2023-10-13 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | up to 2 years
  PFS is defined as the time from D1 of treatment with the study combination until the criteria for disease progression is met as defined by RECIST 1.1 criteria or death as a result of any cause.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | up to 2 years
  ORR will include confirmed complete response (CR) + confirmed partial response (PR) per RECIST 1.1 divided by the number of patients receiving at least one dose of proposed combination.
Number of Participants Experiencing Grade 3 and 4 Toxicities | up to 30 days post-treatment (approximately 6 months on study)
  Grade 3 and 4 toxicities as defined by the NCI Common Terminology Criteria for Adverse Events (version 5.0) (CTCAE v5.0)
Summary of Grade 3 and 4 Toxicities by Count of participants | up to 30 days post-treatment (approximately 6 months on study)
  Grade 3 and 4 toxicities as defined by the NCI Common Terminology Criteria for Adverse Events (version 5.0) (CTCAE v5.0)
Efficacy of irinotecan measured by PFS for patients with and without irinotecan containing regimens | up to 2 years
  PFS will be compared between those subjects who were treated in the last 4 months with an irinotecan containing regimen versus those who were not

CONTACTS AND LOCATIONS:
Overall Officials: Dustin Deming, MD, Principal Investigator — UW Carbone Cancer Center
Locations (1):
- University of Wisconsin Carbone Cancer Center, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No